CLINICAL TRIAL: NCT07109700
Title: A Randomized, Double-blind, Placebo and Active Comparator-controlled Phase 2 Study to Evaluate the Efficacy and Safety of HDM1005 in Subjects With T2DM With Inadequate Glycemic Control After Diet/Exercise or Metformin Therapy
Brief Title: A Study of HDM1005 in Participants With T2DM Not Controlled With Diet/Exercise or Metformin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HDM1005-201
Record Dates: First submitted 2025-07-25; First posted 2025-08-07 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental group: HDM1005 1 (Experimental): HDM1005 administered subcutaneously (SC)
  Interventions: Drug: HDM1005 1
- Experimental group: HDM1005 2 (Experimental): HDM1005 administered SC
  Interventions: Drug: HDM1005 2
- Experimental group: HDM1005 3 (Experimental): HDM1005 administered SC
  Interventions: Drug: HDM1005 3
- Experimental group: HDM1005 4 (Experimental): HDM1005 administered SC
  Interventions: Drug: HDM1005 4
- Placebo group (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- Active Comparator: Dulaglutide (Active Comparator): Dulagutide administered SC
  Interventions: Drug: Dulaglutide 1.5 MG

INTERVENTIONS:
Drug: HDM1005 1 — administered SC, QW, 20 weeks
  Arms: Experimental group: HDM1005 1
Drug: HDM1005 2 — administered SC, QW, 20 weeks
  Arms: Experimental group: HDM1005 2
Drug: HDM1005 3 — administered SC, QW, 20 weeks
  Arms: Experimental group: HDM1005 3
Drug: HDM1005 4 — administered SC, QW, 20 weeks
  Arms: Experimental group: HDM1005 4
Drug: Placebo — administered SC, QW, 20 weeks
  Arms: Placebo group
Drug: Dulaglutide 1.5 MG — administered SC, QW, 20 weeks
  Arms: Active Comparator: Dulaglutide

SUMMARY:
This study is a multicenter, randomized, double-blind (with open-label dose levels and active comparator), parallel-group, placebo- and active-controlled Phase 2 clinical trial aimed at evaluating the efficacy, safety, immunogenicity, and pharmacokinetic (PK) characteristics of HDM1005 in subjects with Type 2 Diabetes Mellitus (T2DM) who have inadequate glycemic control after diet/exercise or metformin therapy.

A total of 216 subjects will be enrolled. All subjects will be stratified by baseline HbA1c levels (≤8.5% or >8.5%) and prior metformin use, then randomized 1:1:1:1:1:1 to: Group 1 (HDM1005 0.5 mg), Group 2 (HDM1005 1.0 mg), Group 3 (HDM1005 2.0 mg), Group 4 (HDM1005 3.0 mg), Group 5 (Placebo), and Group 6 (open-lable dulaglutide 1.5 mg, active comparator), with 36 subjects in each treatment group. Within each dose cohort (0.5/1.0/2.0/3.0mg), there will be ~45 total subjects (36 HDM1005 + 9 placebo). The 1.0mg, 2.0mg, and 3.0mg cohorts will implement dose titration.

The study consists of: 2-week screening, 20-week treatment, and 4-week safety follow-up. The end-of-study visit will be conducted 28 days after the last administration cycle.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed as Type 2 Diabetes Mellitus (T2DM) for at least 24 weeks;
* Hemoglobin A1c (HbA1c) ≥7.5% and ≤10.5%
* Body Mass Index (BMI within the range of 22.5 ~ 40.0 kg/m2

Exclusion Criteria:

* Other types of diabetes besides T2DM
* Acute complications of diabetes (such as diabetic ketoacidosis, diabetic lactic acidosis, or hyperosmolar non-ketotic coma) occurred within 24 weeks prior to signing the Informed Consent Form (ICF)
* History of a level 3 hypoglycemic episode or a history of asymptomatic hyp oglycemic episodes within 24 weeks prior to signing the ICF
* History or family history of medullary thyroid carcinoma (MTC), thyroid C-cell hyperplasia, or multiple endocrine neoplasia type 2 (MEN2)
* History of acute or chronic pancreatitis; or presence of risk factors for pancreatitis; or history of symptomatic gallbladder disease within 24 weeks prior to signing the ICF
* Investigator determines that the subject has a condition or disease affecting gastric emptying or gastrointestinal nutrient absorption, such as weight-loss surgery or other gastric resections, irritable bowel syndrome, dyspepsia, or gastroparesis
* Use of antidiabetic medications within 12 weeks prior to signing the ICF
* Hemoglobin (Hb) <100 g/L (female) or <110 g/L (male)
* FPG ≥13.9 mmol/L
* Aspartate aminotransferase (AST) >2.5× upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >2.5× ULN
* Total bilirubin >1.5× ULN
* Fasting triglyceride (TG) >5.6 mmol/L (500 mg/dL)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 20
  HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.

SECONDARY OUTCOMES:
Change from baseline in HbA1c | Baseline, Week 12
  HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
The percentage of patients reaching the HbA1c target of ≤6.5% and of ≤7.0% | Week 20
  HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Change frome baseline in fasting plasma glucose (FPG) | Baseline, Week 12 and Week 20
  FPG is a test to determine sugar levels in serum sample after an overnight fast.
Change from baseline in body weight | Baseline, Week 12 and Week 20
  Change from baseline in body weight is calculated by subtracting the baseline weight measurement from the post-treatment weight measurement at a specified time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No